CLINICAL TRIAL: NCT02678468
Title: Early Vision Screening With Automated Photorefraction in Pre-term, Low-birth- Weight and Development-delay Children in Far-Eastern Memorial Hospital, Taiwan
Brief Title: Early Vision Screening in High-risk Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yao-Lin Liu, M.D., Far Eastern Memorial Hospital
Other Study IDs: 104077-F
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Amblyopia; Child
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- high-risk group: children with birth history of pre-term, low birth weight children with develop delay
- normal group: children with normal birth history and normal development

SUMMARY:
To evaluate the effect of early vision screening with automated photorefraction device in high risk children

DETAILED DESCRIPTION:
Pre-term, low-birth-weight, and development delay are well-known risk factors related to higher incidence of high refractive error and strabismus, which can potentially lead to amblyopia and is regarded as amblyopia risk factors. This project is a cross-sectional controlled study. Our study includes high-risk group and normal group. High-risk group includes children with birth history of pre-term, low-birth-weight and the diagnosis of development delay in FEMH. Normal group enrolled age-matched children without those risk factors. Vision screening by FDA-approved photorefraction device as well as comprehensive ophthalmic exams for definite diagnosis will be performed on the high-risk group and the normal group.

ELIGIBILITY:
Inclusion Criteria:

* High risk group: children with gestational age less than 36weeks, birth weight less than 2500g and children diagnosed as develop delay
* Normal group: children with normal birth history and normal development

Exclusion Criteria:

* Children with known ophthalmic diseases
* Children with congenital systemic diseases

Ages: 1 Year to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children born and regular followed at pediatric clinic in Far Eastern Memorial Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
positive predictive value of vision screening | one year
  positive predictive value

SECONDARY OUTCOMES:
Odds ratio of having amblyopia risk factors | one year
  Odds ratio

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Lin Liu, M.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Other, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bloomberg JD, Suh DW. The accuracy of the plusoptiX A08 photoscreener in detecting risk factors for amblyopia in central Iowa. J AAPOS. 2013 Jun;17(3):301-4. doi: 10.1016/j.jaapos.2013.03.014. PMID 23791414